CLINICAL TRIAL: NCT05213845
Title: Assessment of Spine Rehabilitation Program Using Spine Flexion and Extension Full Active Range of Motion for Patients With Chronic Low Back Pain : a Monocentric Prospective Cohort Study
Brief Title: Spine Rehabilitation Using Spine Flexion / Extension Full Active Range of Motion for Patients With Chronic Low Back Pain
Acronym: REACTIVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment to meet the objectives in time
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHR 1206; 2021-A02319-32 (Other: ANSM)
Record Dates: First submitted 2022-01-17; First posted 2022-01-28 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-02

CONDITIONS: Low Back Pain
Keywords: rehabilitation; active range of motion; kinesiophobia; physiotherapy
MeSH Terms: conditions — Low Back Pain; Kinesiophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with chronic low back pain (Other)
  Interventions: Procedure: Spine flexion/extension active range of motion exercises

INTERVENTIONS:
Procedure: Spine flexion/extension active range of motion exercises — Five full active range of motion rehabilitation sessions will be scheduled. Four or the five following full active range of motion exercises will be performed during one rehabilitation session : spine flexion and extension (quadrupedic position), lumbar flexion and extension (sitting position), posterior and anterior pelvic tilt (sitting and standing position), lumbar flexion and extension (standing position) and Jefferson Curl exercise. All five rehabilitation sessions must be performed within 60 days

SUMMARY:
The main objective of this study is to assess efficacy of a spine rehabilitation program, using spine flexion and extension full active range of motion, on physical disability of patients with chronic low back pain.

DETAILED DESCRIPTION:
Secondary objectives

The other objectives of this study are to assess the impact of spine rehabiliation program using spine flexion and extension full active range of motion on :

* pain intensity ;
* kinesiophobia
* active range of motion of lumbar flexion and lumbar extension

Conduct of research

After receiving the written consent of the study, participants will benefit from 5 sessions of spine flexion and extension full active range of motion exercises. The following tests and questionnaires will be performed before (baseline) and after (posttreatment) the 5 sessions :

* Visual Analogue Pain Scale,
* Fear Avoidance Beliefs Questionnaire (FABQ),
* Double-inclinometer to measure active range of motion of lumbar flexion and lumbar extension.

ELIGIBILITY:
Inclusion Criteria:

* Medical prescription for chronic low back pain rehabilitation
* Evolution of low back pain for at least 3 months
* No treatment or rehabilitation for low back pain performed within 12 months before enrollment
* Written informed consent given

Exclusion Criteria:

* Spinal fracture or previous spinal surgery
* Cognitive impairments that prevent from understanding the rehabilitation exercises
* Patient with insufficient understanding or expression in French
* Non-mechanical pain : gradually worsening pain, present at rest and especially at night
* Neurological symptom : deficit in the control of bladder and anal sphincters, motor weakness of lower limbs, Cauda equina syndrome
* Pubis paresthesia (or perineum)
* Severe trauma (such as fall from height, traffic accident)
* Unexplained weight loss
* History of cancer
* Drug use or long-term use of corticosteroid
* Spinal deformity
* Altered general condition
* Patient with signs of neurological impairment : positive Lasegue test (Straight Leg Raise Test) or positive Slump test, or DN4 questionnaire greater than or equal to 4
* Patient suffering from a central or peripheral neurological pathology
* Patient taking a level II (weak opiates) or III (morphine and related substances) analgesic treatment
* Patient under guardianship, curatorship or legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Roland-Morris disability questionnaire | Posttreatment (2 months)
  The Roland-Morris questionnaire is a 24-item self report questionnaire assessing physical disability, ranging from 0 (no disability) to 24 (severe disability).

SECONDARY OUTCOMES:
Pain intensity | Posttreatment (2 months)
  Pain intensity will be measured with a Visual Analog Pain Scale, from 0 (no pain) to 10 (pain of maximum intensity)
Fear Avoidance Beliefs Questionnaire (FABQ) | Posttreatment (2 months)
  The FABQ is a patient reported questionnaire which specifically focuses on how patient's fear-avoidance beliefs about physical activity may affect and contribute to his/her low back pain and resulting disability.
Active range of motion of lumbar flexion and lumbar extension | Posttreatment (2 months)
  Active range of motion of lumbar flexion and lumbar extension will be measured with two inclinometers.

CONTACTS AND LOCATIONS:
Locations (1):
- Cabinet de masso-kinésithérapie, Mulhouse, France

IPD SHARING:
Plan to Share IPD: No